CLINICAL TRIAL: NCT03427086
Title: Safety and Tolerability of High Dose Biotin in Patients With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Johnny Salameh, MD, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIO-2017-0270
Record Dates: First submitted 2018-01-29; First posted 2018-02-09 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; Biotin
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Biotin

STUDY DESIGN:
Intervention Model Description: Prospective, double blind, placebo control, randomized 2:1 study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subjects, care givers, investigator, and coordinator will be blinded. The pharmacist, who will be responsible for the drug supply, will be unblinded. The investigational drug and the placebo will have identical pill shape and color. They will be supplied in identical boxes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional (Active Comparator): Patient will received high dose of biotin (300 mg/day)
  Interventions: Drug: Biotin
- Placebo (Placebo Comparator): Patients will receive placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Biotin — High dose biotin
  Other Names: vitamin B7
  Arms: Interventional
Drug: Placebo Oral Tablet — Placebo tablet similar in shape and size to the biotin tablet
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized double blinded randomized 2:1 study. The duration of the study is 6 month. The safety and tolerability of high doses of biotin (300 mg/ day) will be compared to placebo in patients with amyotrophic lateral sclerosis. Patients will be evaluated at baseline, 3, and 6 month. The primary outcome will be any adverse effects recorded. The secondary outcomes will be motor disability measured by ALS-FRS, change in Pulmonary function test parameters (FEV1- FVC), change in subject weight (in kg).

ELIGIBILITY:
Inclusion Criteria:

* Amyotrophic Lateral Sclerosis (ALS) volunteers must be diagnosed within 3 years prior to participation as having possible, probable, or definite ALS, either sporadic or familial according to modified El Escorial criteria
* Age 18-80, able to provide informed consent, and comply with study procedures
* Participants must not have started Riluzole and/or Nuedexta for at least 30 days, or be on a stable dose of Riluzole and/or Nuedexta for at least 30 days, prior to screening (Riluzole and/or Nuedexta -naïve participants are permitted in the study)

Exclusion Criteria:

* The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the participant to provide informed consent, according to PI judgment.
* Exposure to any experimental agent within 30 days of entry or at any time during the trial or enrollment in another research study within 30 days of or during this trial.
* Slow Vital Capacity test less than 50% of the predicted value Patients who had already undergone tracheostomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 6 months
  Any adverse effects resulting from receiving high dose biotin in patients with amyotrophic lateral sclerosis will be recorded

SECONDARY OUTCOMES:
Motor disability measurement | 6 months
  The motor disability will be measured in the both arms using the revised amyotrophic lateral sclerosis functional rating scale (ALS-FRSr). This scale measures the progression and the severity of the disease. It is compose of 12 questions, each questions can have a score from 0 to 4. Questions 1 to 3 are related to bulbar onset, questions 4 to 9 are related to limb onset and questions 10-12 are related to respiratory onset. The minimum score is 0 and the maximum total score is 48. The higher the score the better the functional status. The lower the score the worse the functional status of the patient.
Change in Pulmonary function test parameters ( FEV1- FVC) | 6 months
  Forced expiratory volume in 1 second (FEV1) measured in percents and forced vital capacity (FVC) measured in liters will be measured in the both study arms.
Weight changes | 6 months
  Changes in body weight (in kilograms) will be measured in both study arms

CONTACTS AND LOCATIONS:
Overall Officials: Achraf Makki, MD, Principal Investigator — American University of Beirut Medical Center; Johnny Salameh, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American univeristy of Beirut medical center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kawamata H, Manfredi G. Mitochondrial dysfunction and intracellular calcium dysregulation in ALS. Mech Ageing Dev. 2010 Jul-Aug;131(7-8):517-26. doi: 10.1016/j.mad.2010.05.003. Epub 2010 May 20. PMID 20493207
- [Result] Wijesekera LC, Leigh PN. Amyotrophic lateral sclerosis. Orphanet J Rare Dis. 2009 Feb 3;4:3. doi: 10.1186/1750-1172-4-3. PMID 19192301
- [Result] Musaro A. Understanding ALS: new therapeutic approaches. FEBS J. 2013 Sep;280(17):4315-22. doi: 10.1111/febs.12087. Epub 2013 Jan 3. PMID 23217177
- [Result] Zimmermann KC, Bonzon C, Green DR. The machinery of programmed cell death. Pharmacol Ther. 2001 Oct;92(1):57-70. doi: 10.1016/s0163-7258(01)00159-0. PMID 11750036
- [Result] Celsi F, Pizzo P, Brini M, Leo S, Fotino C, Pinton P, Rizzuto R. Mitochondria, calcium and cell death: a deadly triad in neurodegeneration. Biochim Biophys Acta. 2009 May;1787(5):335-44. doi: 10.1016/j.bbabio.2009.02.021. Epub 2009 Mar 4. PMID 19268425
- [Result] Atamna H, Newberry J, Erlitzki R, Schultz CS, Ames BN. Biotin deficiency inhibits heme synthesis and impairs mitochondria in human lung fibroblasts. J Nutr. 2007 Jan;137(1):25-30. doi: 10.1093/jn/137.1.25. PMID 17182796
- [Result] Stys PK, Zamponi GW, van Minnen J, Geurts JJ. Will the real multiple sclerosis please stand up? Nat Rev Neurosci. 2012 Jun 20;13(7):507-14. doi: 10.1038/nrn3275. PMID 22714021
- [Result] Luessi F, Siffrin V, Zipp F. Neurodegeneration in multiple sclerosis: novel treatment strategies. Expert Rev Neurother. 2012 Sep;12(9):1061-76; quiz 1077. doi: 10.1586/ern.12.59. PMID 23039386
- [Result] Sedel F, Papeix C, Bellanger A, Touitou V, Lebrun-Frenay C, Galanaud D, Gout O, Lyon-Caen O, Tourbah A. High doses of biotin in chronic progressive multiple sclerosis: a pilot study. Mult Scler Relat Disord. 2015 Mar;4(2):159-69. doi: 10.1016/j.msard.2015.01.005. Epub 2015 Jan 24. PMID 25787192
- [Result] Tourbah A, Lebrun-Frenay C, Edan G, Clanet M, Papeix C, Vukusic S, De Seze J, Debouverie M, Gout O, Clavelou P, Defer G, Laplaud DA, Moreau T, Labauge P, Brochet B, Sedel F, Pelletier J; MS-SPI study group. MD1003 (high-dose biotin) for the treatment of progressive multiple sclerosis: A randomised, double-blind, placebo-controlled study. Mult Scler. 2016 Nov;22(13):1719-1731. doi: 10.1177/1352458516667568. Epub 2016 Sep 1. PMID 27589059
- See also: Circulation and Energy Metabolism of the Brain — https://www.ncbi.nlm.nih.gov/books/NBK20413/